CLINICAL TRIAL: NCT03116737
Title: Phase III, Multicenter, Randomized, Double-Blind, Placebo- Controlled Parallel-Designed Evaluation to Assess Safety and Efficacy of Topical Benzocaine for Treatment of Pain Associated With Acute Otitis Media in Children Ages 5 to 12 Years
Brief Title: Phase III Study Evaluating Topical Benzocaine for Treatment of Acute Otitis Media in Children
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Lachlan Pharma Holdings (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LP7700
Record Dates: First submitted 2017-04-03; First posted 2017-04-17 (Actual); Last update posted 2017-10-13 (Actual); Status verified 2017-10

CONDITIONS: Pain; Acute Otitis Media
Keywords: AOM
MeSH Terms: conditions — Pain; Otitis Media

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Benzocaine Otic Solution (Experimental)
  Interventions: Drug: Benzocaine Otic Solution
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Benzocaine Otic Solution
  Arms: Benzocaine Otic Solution
Drug: Placebo
  Other Names: Topical otic solution
  Arms: Placebo

SUMMARY:
The Phase III study is designed to assess the safety, tolerability, and efficacy of Topical Benzocaine in children, ages 5 to 12 years, presenting with Acute Otitis Media-associated ear pain.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients ages 5 to 12 years of age with a clinical diagnosis of unilateral AOM, and with ear pain (current episode <2 weeks duration). Baseline pain entry requires a minimum score of 4 on the FPS-R.
* Patients/guardians must provide Institutional Review Board (IRB) approved written assent, as appropriate, which must be accompanied by an IRB approved written informed consent form (ICF) from the patient's legally acceptable representative (i.e., parent or guardian), as applicable. In addition, all patients or their legally acceptable representatives (i.e., parent or guardian) must sign a Health Insurance Portability and Accountability Act (HIPAA) authorization, if applicable.
* Patients must be physically active and otherwise judged to be in good health on the basis of the medical history and a limited physical examination, as determined by the Investigator.
* Females of childbearing potential must also have a negative urine human chorionic gonadotropin (hCG) pregnancy test on the Study Day, Visit 1.

Exclusion Criteria:

* Patients unable or refusing to independently and consistently complete the FPS-R pain measurements.
* Patients with bilateral AOM, perforated tympanic membrane, history of a perforated tympanic membrane in the last 6 months, or if a perforated tympanic membrane could not be ruled out by speculum examination, impedance testing tympanometry, pneumatic otoscopy, or a Valsalva maneuver.
* Patients who are subsequently diagnosed with a perforated membrane during treatment are to be discontinued immediately.
* Patients with indwelling tympanostomy tubes or draining otitis in the affected ear(s), bullous lesions, erythema of the tympanic membrane without other evidence of AOM, and patients with an anatomic defect of the ear or nasopharynx.
* Complications of treated/untreated ear disease other than qualifying AOM over the past 2 weeks.
* Patients with comorbidity requiring antibiotic therapy, allergy to study medication, immunologic deficiency, and major medical condition(s).
* Patients presenting with methemoglobinemia or a history of methemoglobinemia, vertigo, inherited enzyme deficiencies (including G6PD), impaired cardiac or respiratory functions, epilepsy, heart diseases, hypersensitivity to benzocaine or any other related drug product, inflamed or infected skin, dermatitis, previous medication related shock episode, hepatic impairment, or myasthenia gravis.
* Acute or chronic otitis externa.
* Chronic otitis media (current episode ≥ 2 weeks).
* Patients who smoke.
* Dermatitis involving the affected external ear canal or pinna.
* Any topical or systemic antibiotic received within the 14 days prior to study entry.
* Patients administered vaccinations a week prior to or on any of the Study Day Visits.
* Any ear drops, topical drying agent or over-the-counter (OTC) therapy for any ear related issue received within 36 hours prior to enrollment.
* Fever >102°F or at any elevated level considered necessary by the study investigator.
* Known hypersensitivity to the study drug or similar compounds including any of the inactive ingredients.
* Patients receiving medication on a chronic basis for pain (including steroidal or non-steroidal anti-inflammatory drugs).
* Oral analgesics such as ibuprofen/acetaminophen within 6 hours prior to study entry.
* Use of drug products with potential interactions including sulfonamides, aminosalicylates, anti-cholinesterases, suxamethonium, antiarrhythmics, monoamine oxidase inhibitors, or tricyclic antidepressants within 14 days.
* Eating, drinking, chewing of gum, or use of mints/lozenges during the first hour after initial study dose.
* Children that use pacifiers and/or are still breastfed.
* Exposure to any investigational agent within the 30 days prior to study entry.
* Previous enrollment in this study.
* Pregnant or lactating.
* Clinically significant mental or emotional illnesses (by history or as determined by the on-site investigator).
* The child has a condition or demonstrates a behavior that the Investigator or site personnel believe would interfere with the ability to provide assent (age appropriate) or comply with study instructions/tasks, or that might confound the interpretation of the study results, or put the child or others at risk.

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 141 (Actual)
Dates: Start 2017-01-03 (Actual); Primary Completion 2017-07-21 (Actual); Study Completion 2017-07-21 (Actual)

PRIMARY OUTCOMES:
Summed Pain Intensity Difference Assessed by Faces Pain Scale-Revised (FPS-R) | 60 minutes

SECONDARY OUTCOMES:
Summed Pain Intensity Difference Assessed by Faces Pain Scale-Revised (FPS-R) | 120 minutes
Pain Intensity Difference Assessed by Faces Pain Scale-Revised (FPS-R) | Up to 3 days
Dosing Intervals | Up to 3 days
Use of Rescue Medications | Up to 3 days
Assess the Safety and Tolerability of Benzocaine Based on Reported Adverse Events | Up to 3 days
  Safety will be assessed by adverse event reporting on all study days. Fisher's exact test will be used to compare adverse event rates between treatment groups for the following categories: 1) all adverse events; 2) treatment related adverse events; 3) severe adverse events; 4) serious adverse events; 5) discontinuation due to adverse event.
Assess the Safety and Tolerability of Benzocaine Based on Physical Examinations | Up to 3 days
  Physical examinations will be assessed. For each body system of the physical examination, the shift from normal/abnormal will be presented by treatment group as the number and percentage of children.
Assess the Safety and Tolerability of Benzocaine Based on Vital Signs | Up to 3 days
  Vital signs (blood pressure, pulse, temperature, and respiratory rate) will be assessed. Descriptive statistics will be presented for the vital signs measurements collected, as well as the vital sign changes from Day 1 to Day 3 by treatment group.

CONTACTS AND LOCATIONS:
Locations (1):
- Cyn3rgy Research, Gresham, Oregon, United States

IPD SHARING:
Plan to Share IPD: No